CLINICAL TRIAL: NCT01954004
Title: An Open Registry to Measure the Impact of Adding Genomic Testing (Prolaris®) on the Treatment Decision Following Biopsy in Newly Diagnosed Prostate Cancer Patients
Brief Title: Open Registry Measuring Impact of Genomic Testing on Treatment of Prostate Cancer Patients
Status: Completed | Type: Observational
Sponsor: Myriad Genetic Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PROCEDE-1000
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
This registry is intended to evaluate the impact of genomic test results towards selecting a first-line therapy option for newly diagnosed localized prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed (≤6 months), untreated patients with histologically proven adenocarcinoma of the prostate that have the following characteristics.
* Clinically localized (no evidence on clinical or imaging studies of advanced disease).
* No hormonal therapy including LHRH (luteinizing hormone-releasing hormone) agonist or antagonist, anti-androgen, estrogens or exogenous androgens, when applicable.
* Sufficient amount of tissue remains from biopsy to perform genomic testing.

Exclusion Criteria:

* Patients with a known history of hypogonadism

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recently diagnosed treatment-naïve patients with early stage localized prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 1270 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Percentage change from the recorded PRE-Prolaris® test treatment option versus the ACTUAL treatment option implemented following results of genomic risk assessment testing (Prolaris®). | 4 months

SECONDARY OUTCOMES:
Percentage change from the recorded PRE-Prolaris® test treatment option versus the POST-Prolaris® test treatment plan following review of the genomic test results (prior to patient consultation) | 1 month
Percentage change from the recorded PRE-Prolaris® test treatment option versus the POST-Prolaris® test treatment plan following consultation with the patient. | 2 months

OTHER OUTCOMES:
• The mean change in the physician's likelihood of recommending non-interventional therapy (watchful waiting or active surveillance) post-genomic testing compared to pre-genomic testing. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Wenstrup, MD, Study Director — Myriad Genetic Laboratories, Inc.
Locations (1):
- Salt Lake City, Utah, United States